CLINICAL TRIAL: NCT06077968
Title: Retrospective Study Evaluating ABRYSVO Vaccine Effectiveness Against Severe Lower Respiratory Tract Infection in Older Adults
Brief Title: A Study to Learn About ABRYSVO Vaccine in Older Adults to Prevent Severe Respiratory Syncytial Virus (RSV) Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: C3671030; NCT06077968 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Viruses
Keywords: Lower respiratory tract infections; Acute respiratory infections; vaccine; RSV vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Standard of care specimens will be salvaged and tested on a multiplex respiratory panel at a contracted vendor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccinated: Patients will be considered vaccinated if they have documented evidence of receiving ABRYSVO ≥21 days before index date (i.e., defined as the date of hospitalization or Emergency Department (ED) admission.)
  Interventions: Biological: Prior standard of care receipt of Pfizer's ABRYSVO vaccine
- Unvaccinated: Patients will be considered unvaccinated if they do not have documented evidence of receiving ABRYSVO.
  Interventions: Biological: Prior standard of care receipt of Pfizer's ABRYSVO vaccine

INTERVENTIONS:
Biological: Prior standard of care receipt of Pfizer's ABRYSVO vaccine — Participants will receive Pfizer's ABRYSVO vaccine as part of standard of care. Vaccine is not administered in this study.

SUMMARY:
The main purpose of this study is to learn about the effectiveness of Pfizer's ABRYSVO vaccine. This vaccine helps to prevent infections caused by Respiratory Syncytial Virus (RSV). RSV is a virus that can cause infections in the airways. These symptoms can be cold-like symptoms, but in some cases can lead to severe symptoms or hospitalization.

This study uses only healthcare data that are already collected from routine visits to healthcare providers. This means that participants will not be actively enrolled in the study and there are no study treatments. The study will look at data for about two years. This study will look at patient information from:

* Adults ages 60 years and older
* Adults who are eligible to receive the ABRYSVO vaccination

Substudy A:

* This study will assess the duration of protection of ABRYSVO in adults ages 60 years and older after completion of the original study.
* The substudy will look at data from subsequent RSV seasons after the first dose of ABRYSVO for about 3 years.

Substudy B:

* This study will assess vaccine effectiveness of ABRYSVO after revaccination in routine use, pending ACIP recommendation for revaccination.
* The substudy will look at data for about 2 years after revaccination.

DETAILED DESCRIPTION:
The overall research question asks how effective ABRYSVO® is against severe RSV disease in real-world populations. The primary objective of this study is to estimate the VE of Pfizer's ABRYSVO® vaccine against RSV-related LRTD hospitalizations among Kaiser Permanente Southern California members who are eligible for vaccination per current Advisory Committee on Immunization Practices (ACIP) recommendations. Key secondary objectives include determining ABRYSVO® VE against RSV-related LRTD hospitalizations among the immunocompetent and stratified by age group (60-74 years vs 75 years and older). Additional secondary objectives include assessment of ABRYSVO® VE stratified by RSV subgroup, against ARI endpoints, death, among high-risk subgroups, and against critical outcomes.

A case control study with test negative design will be the primary analysis assessing RSV-related outcomes. An exploratory cohort design may also be used to assess all-cause outcomes and RSV-related outcomes.

Standard-of-care specimens (e.g. stored remnant respiratory specimens) from patients who did not receive RSV testing, who tested negative for RSV via RSV-only test, or a had limited multiplex viral respiratory panel assay will be salvaged and tested using a full respiratory multiplex polymerase chain reaction (PCR) panel at KPSC. Further, all RSV positives will be tested for RSV A and RSV B.

ELIGIBILITY:
Inclusion Criteria:

1. KPSC patients eligible to receive ABRYSVO® per current ACIP recommendations for adults ages 60 and older who are admitted to the hospital with ARI/LRTD, (defined using International Classification of Diseases (ICD) codes after start of study period, and who have had an RSV test, either through SOC testing or blinded study testing of remnant respiratory specimens.
2. For secondary objectives estimating VE against ED admission, the TND will include KPSC patients eligible to receive ABRYSVO® who present to the ED with ARI/LRTD after start of study period, and who have had an RSV test, either through standard of care testing or blinded study testing of remnant respiratory specimens.
3. For exploratory objectives estimating VE against RSV-related cardiac hospitalization, the TND will include KPSC patients eligible to receive ABRYSVO® who are hospitalized or present to the ED with cardiac events (defined using ICD codes) after start of study period, and who have had an RSV test, either through SOC testing or blinded study testing of remnant respiratory specimens.
4. We will include membership requirement of 1 year prior to index date, which is defined as the date of hospitalization or ED admission (allowing 45-day administrative gap), to facilitate accurate capture of comorbid conditions.

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

We will exclude patients who receive another licensed or investigational RSV vaccine prior to hospitalization or ED visit from the study population and analysis. Patients will be excluded if the index date is within certain time windows from vaccination date, outlined further in the exposure section below.

SSA and SSB Eligibility Criteria:

The inclusion criteria for Substudy A are described above for the Test Negative Design.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective database study using existing healthcare data, no patients will be actively enrolled.
  This study will be conducted at KPSC, an integrated health care organization comprising one of the largest health insurance plans in the United States (US), a hospital system, and >7,800 physicians and 27,000 nurses located throughout 9 counties of Southern California. Approximately half of the KPSC network will be included in this study. For the TND, the study population will include all KPSC patients eligible for vaccination ages 60 and older per current ACIP recommendations who are admitted to the hospital or present to the ED with ARI or LRTD or cardiac events (exploratory objective) after study start, and who have had a respiratory specimen collected with an RSV test result, either through SOC testing or study testing of remnant SOC specimens.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
1. Vaccine Effectiveness (VE) calculated as 1 minus the odds ratio (OR) comparing the odds of being vaccinated with ABRYSVO for RSV-related hospitalized LRTD cases and controls, multiplied by 100%. | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO against RSV-related LRTD hospitalizations

SECONDARY OUTCOMES:
Key Secondary 1: Among the immunocompetent, VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related LRTD hospitalizations cases and controls, multiplied by 100%. | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations among the immunocompetent.
Key Secondary 2: ABRYSVO® VE estimates stratified by age group | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations stratified by age group (60-74 years vs 75 years and older)
Secondary 3: To further describe the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations stratified by RSV subgroup (A and B) | Up to 2 years
  Adjusted for confounding factors using logistic regression. ABRYSVO® VE estimates stratified by virus subgroups
Secondary 4: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related severe LRTD cases and controls, multiplied by 100% | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related severe LRTD.
Secondary 5: ABRYSVO® VE estimates stratified by frailty index | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalization stratified by frailty index.
Secondary 6: ABRYSVO® VE estimates stratified by chronic medical condition risk category | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations, stratified by chronic medical condition risk category (3 strata: not high-risk conditions, immunocompromising high-risk conditions, non-immunocompromising high-risk conditions).
Secondary 7: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized LRTD cases and controls, multiplied by 100%, among those with CHF or COPD | Up to 2 years
  Adjusted for confounding factors using logistic regression. Among those with congestive heart failure (CHF) or Chronic Obstructive Pulmonary Disease (COPD,) to estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations
Secondary 8-1: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for ED (without subsequent hospitalization) cases and controls, multiplied by 100% | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against ED admission (without subsequent hospitalization)
Secondary 8-2: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for hospitalized or ED visit (without subsequent hospitalization) cases and controls, multiplied by 100%. | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against ED (without subsequent hospitalization) or hospitalization
Secondary 9: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related death cases and controls, multiplied by 100%. | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related death
Secondary 10-1: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for hospitalized RSV-related ARI cases and controls, multiplied by 100% | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related ARI hospitalization
Secondary 10-2: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related ARI ED visit (without subsequent hospitalization) cases and controls, multiplied by 100% | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related ARI ED visits (without subsequent hospitalization).
TND Secondary 10-3: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for ED visit (without subsequent hospitalization) or hospitalized RSV-related ARI cases and controls, multiplied by 100% | 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related hospitalization or ED visits (without subsequent hospitalization)
TND Secondary 11: Describe age, sex, race/ethnicity, clinical and laboratory characteristics, and disease severity (length of stay [LOS], intensive care unit [ICU] admission, respiratory support) of any patients who received ABRYSVO | Up to 2 years
  To describe demographic, clinical, and laboratory characteristics and disease severity of any RSV events among vaccinated individuals as compared to unvaccinated
Secondary 12: ABRYSVO® RSV-related VE estimates stratified by age group and chronic medical risk categories | Up to 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations stratified by age group and chronic medical risk categories.
Secondary 13: ABRYSVO® VE estimates stratified by immunocompromised status | 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations stratified by (1) immunocompromised vs immunocompetent, and separately (2) within those with immunocompromising condition, by severe vs moderate immunocompromised status.
Secondary 14: VE calculated as 1 minus the odds ratio (OR) comparing the odds of being vaccinated with ABRYSVO® for hMPV-related hospitalized ARI/LRTD cases and controls, multiplied by 100% | 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against hMPV-related ARI/LRTD hospitalizations
Secondary 15: ABRYSVO® VE estimates stratified by age group. | 2 years
  Adjusted for confounding factors using logistic regression. To estimate ABRYSVO® VE against RSV-related LRTD hospitalizations by alternative age groups 60-69 years, 70-79 years, 80 years and older
Secondary 16: Among the immunocompetent, VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized/ED visits LRTD cases and controls, multiplied by 100% | 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) among the immunocompetent.
Secondary 17: ABRYSVO® VE estimates stratified by age group | 2 years
  Adjusted for confounding factors using logistic regression. To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization), stratified by age group (60-74 years vs 75 years and older)
SSA Primary: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100%, using LRTD events from the 3rd season | Up to 3 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) during the 3rd RSV season after a single dose
SSA Secondary 1: VE calculated as 1 minus the OR comparing the odds of ABRYSVO® vaccination and timing compared with unvaccinated, stratified by time since vaccination, multiplied by 100%, using LRTD hospitalization/ED events from the 3rd season | Up to 3 years
  To estimate effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) in the third season after a single dose by time since vaccination, defined in 3-month intervals up to 36 months
SSA Secondary 2: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100%*, using LRTD events from the 2nd season | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) during the 2nd RSV season after a single dose
SSA Secondary 3: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100%, using LRTD events from the 4th season | Up to 4 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) during the 4th RSV season after a single dose
SSA Secondary 4: VE calculated as 1 minus the OR comparing the odds of being vaccinated with ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100%*, using LRTD events from the 5th season | Up to 5 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED visits (without subsequent hospitalization) during the 5th RSV season after a single dose
SSA Secondary 5: VE calculated as 1 minus the OR comparing the odds of ABRYSVO® vaccination and timing compared with unvaccinated, stratified by time since vaccination, multiplied by 100%, using LRTD hospitalization/ED events from the 2nd season | Up to 2 years
  To estimate effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations/ED visits (without subsequent hospitalization) in the second season after a single dose by time since vaccination, defined in 3-month intervals up to 24 months
SSA Secondary 6: VE calculated as 1 minus the OR comparing the odds of ABRYSVO® vaccination and timing compared with unvaccinated, stratified by time since vaccination, multiplied by 100%, using LRTD hospitalization/ED events from the 4th season | Up to 4 years
  To estimate effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations/ED visits (without subsequent hospitalization) in the fourth season after a single dose by time since vaccination, defined in 3-month intervals up to 48 months
SSA Secondary 7: VE calculated as 1 minus the OR comparing the odds of ABRYSVO® vaccination and timing compared with unvaccinated, stratified by time since vaccination, multiplied by 100%, using LRTD hospitalization/ED events from the 5th season | Up to 3 years
  To estimate effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations/ED visits (without subsequent hospitalization) in the fifth season after a single dose by time since vaccination, defined in 3-month intervals up to 60 months
SSB Primary: VE calculated as 1 minus the odds ratio comparing the odds of being vaccinated with two doses of ABRYSVO® vs not vaccinated with any dose of ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100% | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED events (without subsequent hospitalization) after revaccination among those with 2 vs 0 dose of ABRYSVO®, in the first season after revaccination
SSB Secondary 1: VE calculated as 1 minus the OR comparing the odds of being vaccinated with two doses of ABRYSVO® vs being vaccinated with one dose of ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100% | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED events (without subsequent hospitalization) after revaccination among those with 2 vs 1 dose of ABRYSVO®, in the first season after revaccination
SSB Secondary 2: VE calculated as 1 minus the OR comparing the odds of being vaccinated with two doses of ABRYSVO® vs not vaccinated with any dose of ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100% | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED events (without subsequent hospitalization) after revaccination among those with 2 vs 0 dose of ABRYSVO®, in the second season after revaccination
SSB Secondary 3: VE calculated as 1 minus the OR comparing the odds of being vaccinated with two doses of ABRYSVO® vs being vaccinated with one dose of ABRYSVO® for RSV-related hospitalized/ED visit LRTD cases and controls, multiplied by 100% | Up to 2 years
  To estimate the effectiveness of ABRYSVO® against RSV-related LRTD hospitalizations or ED events (without subsequent hospitalization) after revaccination among those with 2 vs 1 dose of ABRYSVO®, in the second season after revaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671030